CLINICAL TRIAL: NCT00960206
Title: Post-Approval Study of the ABC and Trident® Systems
Brief Title: ABC/Trident® Ceramic Post Approval Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stryker Orthopaedics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 33/45
Record Dates: First submitted 2009-08-05; First posted 2009-08-17 (Estimated); Results first posted 2014-08-15 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2016-12

CONDITIONS: Arthroplasty, Replacement, Hip

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Trident®System (Experimental): Trident® Ceramic Insert/Trident® AD HA Acetabular Shell
  Interventions: Device: Trident® Ceramic Insert/Trident® AD HA Acetabular Shell
- ABC System (Experimental): Alumina Insert/PSL® Microstructured Acetabular Shell or Secur-Fit® HA PSL® Acetabular Shell
  Interventions: Device: Alumina Insert/PSL® Microstructured Acetabular Shell or Secur-Fit® HA PSL® Acetabular Shell
- Control (Active Comparator): OmniFit® Series II Insert/OmniFit® PSL® Microstructured Acetabular Shell
  Interventions: Device: OmniFit® Series II Insert/OmniFit® PSL® Microstructured Acetabular Shell

INTERVENTIONS:
Device: Trident® Ceramic Insert/Trident® AD HA Acetabular Shell — Trident® Ceramic Insert/Trident® AD HA Acetabular Shell
  Arms: Trident®System
Device: Alumina Insert/PSL® Microstructured Acetabular Shell or Secur-Fit® HA PSL® Acetabular Shell — Alumina Insert/PSL® Microstructured Acetabular Shell or Secur-Fit® HA PSL® Acetabular Shell
  Arms: ABC System
Device: OmniFit® Series II Insert/OmniFit® PSL® Microstructured Acetabular Shell — OmniFit® Series II Insert/OmniFit® PSL® Microstructured Acetabular Shell
  Arms: Control

SUMMARY:
The purpose of the Post Approval Study of the ABC and Trident® systems is to continue to demonstrate the safety and efficacy of the alumina-on-alumina bearing surfaces combined with the appropriate shell in a cementless application.

DETAILED DESCRIPTION:
The ABC/ Trident® study was initiated in 1996 as an FDA IDE pre-market study in the United States for alumina bearing THR. PreMarket Approval (PMA)application was approved in February 3,2003. The Post Approval Study (PAS) involved six surgeon investigators from the original IDE study. Subjects who consented to participate in the Post Approval Study continued to be followed to collect limited patient reported data regarding status of the hip.

ELIGIBILITY:
Inclusion Criteria:

* The individual has signed a Patient Informed Consent (PIC), specific to this study, and approved by the Institutional Review Board (IRB).
* The individual is between the ages of 21 and 75 years.
* The individual is not classified as morbidly obese.
* The individual clinically qualifies for total hip arthroplastic surgery based on physical examination and medical history.
* The individual is diagnosed with a primary diagnosis of Non-Inflammatory Degenerative Joint Disease (osteoarthritis, traumatic arthritis, avascular necrosis, slipped capital epiphysis, pelvic fracture, femoral fracture, failed fracture fixation or diastrophic variant).
* The individual does not have an active infection within the affected hip joint.
* The individual has not had a previous total hip replacement or hip fusion to the affected hip joint.
* The individual is physically and mentally willing and able to comply with postoperative scheduled clinical and radiographic evaluations and rehabilitation (i.e., not currently being treated for a psychiatric disorder, senile dementia, Alzheimer's disease, presence of alcohol or substance abuse).
* The individual does not have a neuromuscular or neurosensory deficiency that limits the ability to evaluate the safety and effectiveness of the device.
* The individual does not have a diagnosed systemic disease that would affect the subject's welfare or overall outcome of the study (i.e., moderate to severe osteoporosis, Paget's disease, renal osteodystrophy), is not immunologically suppressed, nor receiving steroids in excess of physiologic dose requirements.
* The individual is skeletally mature.
* The individual is not pregnant.
* The individual is not a prisoner.
* The individual has no plans to relocate to another geographic area before the completion of the study.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 413 (Actual)
Dates: Start 2003-03; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Capello, MD, Study Chair — Indiana University School of Medicine; Benjamin Bierbaum, MD, Principal Investigator — New England Baptist Hospital; James D'Antonio, MD, Study Chair — Greater Pittsburgh Orthopaedic Associates; James Roberson, MD, Principal Investigator — Emory Orthopaedics Center; Scott Siverhus, MD, Principal Investigator — Toledo Joint Replacement and Orthopedic Center; Robert Zann, MD, Principal Investigator — Orthopaedic Surgery Associates
Locations (6):
- United States (6):
  - Orthopaedic Surgery Associates, Boca Raton, Florida
  - Emory Univeristy, Atlanta, Georgia
  - Indiana University, Indianapolis, Indiana
  - New England Baptist Hospital, Boston, Massachusetts
  - Toledo Joint Replacement and Orthopedic Center, Toledo, Ohio
  - Greater Pittsburgh Orthopaedics Assoc., Moon Township, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were 413/464 participants/hips enrolled. Started, completed and not completed counts are reported by hip.
Groups:
- Trident® System: Hip received the Trident® Acetabular System with a ceramic insert and ceramic femoral head.
- ABC System: Hip received the ABC Acetabular System with a ceramic insert and ceramic femoral head.
- Control: Hip received the Omnifit Acetabular system with polyethylene insert and metal femoral head.
Period: Overall Study
Arm/Group | Trident® System | ABC System | Control
Started | 190 | 185 | 89
Completed | 150 | 158 | 77
Not Completed | 40 | 27 | 12
Not completed — Death | 7 | 4 | 1
Not completed — Unwilling/Unable to return | 1 | 2 | 0
Not completed — Lost to Follow-up | 8 | 14 | 8
Not completed — Withdrawal by Subject | 2 | 4 | 0
Not completed — Revision of study component | 2 | 2 | 2
Not completed — Missing 10 year data | 20 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are reported by hip for each arm.
Groups:
- Trident System: Trident Ceramic Insert/Trident AD with PureFix HA Shell
- ABC System: Howmedica Osteonics Alumina Insert/either PSL Microstructured or Secur Fit HA PSL Shell
- Control: Howmedica Osteonics Omnifit Series II Cup Inserts/Omnifit PSL Microstructured Shell
- Total: Total of all reporting groups
Arm/Group | Trident System | ABC System | Control | Total
Number analyzed (Participants) | 190 | 185 | 89 | 464
Age, Continuous [Mean (Full Range); unit: years] — An approved protocol deviation allowed enrollment of a 12 y.o. female with juvenile RA.
  years | 51.5 [12 to 74] | 53.9 [26 to 75] | 54.7 [26 to 75] | 53.08 [12 to 75]
Sex/Gender, Customized [Number; unit: hips]
  Female | 67 | 64 | 35 | 166
  Male | 123 | 121 | 54 | 298
Region of Enrollment [Number; unit: hips]
  United States | 190 | 185 | 89 | 464

OUTCOME MEASURES:

1. Primary Outcome: Component Revision and Complications
Description: The number of hips in which the study device was removed and replaced with a new component/s is listed. Complications (adverse events) are listed in the adverse event section.
Time Frame: 10 years
Population: Number of participants analyzed includes all subjects enrolled.
Measure: Number; unit: hips
Units Other Than Participants: hips
Groups:
- Control: Hip recevied the Omnifit Acetabular system with polyethylene insert and metal femoral head.
Arm/Group | Trident® System | ABC System | Control
Number analyzed (Participants) | 177 | 166 | 87
Number analyzed (hips) | 190 | 185 | 89
hips | 2 | 2 | 2
Statistical Analysis 1: Comparison: ABC System vs Control; To compare the Kaplan-Meier survivorship between the two systems; Test type: Superiority or Other; p = 0.0832, Log Rank
Statistical Analysis 2: Comparison: Trident® System vs Control; To compare the Kaplan-Meier survivorship between the two systems; Test type: Superiority or Other; p = 0.1657, Log Rank

2. Secondary Outcome: Harris Hip Score
Description: Scores can range from 0 to 100 with 0 being the worst and 100 being the best score. A score of 80-100 is considered good-excellent and a score less than or equal to 79 is considered fair-poor.
  90 - 100 = excellent
  80 - 89 = good
  70 - 79 = fair
  0 - 69 = poor
Time Frame: 3-5 and 10 Years
Population: Participants may have one or both hips replaced. Number of participants and hips analyzed include all enrolled. Number of hips with HHS evaluated at postoperative periods indicated is included in the outcome results posting.
Measure: Number; unit: hips
Units Other Than Participants: Hips
Arm/Group | Trident® System | ABC System | Control
Number analyzed (Participants) | 177 | 166 | 87
Number analyzed (Hips) | 190 | 185 | 89
hips
  3 yr hips with good-excellent score (80-100) | 160 | 171 | 81
  3 yr hips with a fair-poor score (0-79) | 2 | 2 | 2
  4 yr hips with a good-excellent score (80-100) | 148 | 164 | 77
  4 yr hips with a fair-poor score (0-79) | 6 | 2 | 2
  5 yr hips with a good-excellent score (80-100) | 126 | 158 | 76
  5 yr hips with a fair-poor score (0-79) | 6 | 4 | 2
  10 yr hips with a good-excellent score (80-100) | 67 | 115 | 56
  10 yr hips with a fair-poor score (0-79) | 0 | 4 | 2
Statistical Analysis 1: Comparison: Trident® System vs ABC System vs Control; To compare the # of cases at 10 years for those that have a HHS ≥ 80 to those that have < 80 for all three arms; Test type: Superiority or Other; p = 0.3701, Fisher Exact

3. Secondary Outcome: Radiographic Evaluation
Description: Failure is defined as progressive femoral radiolucency (RLL) > or = 2mm around entire stem, progressive subsidence > or = 5mm, progressive acetabular radiolucency (RLL) > or = 2 mm around entire cup, or cup migration > or = 3mm.
Time Frame: 3-5 and 10 years
Population: Participants may have one or both hips replaced. Number of participants/hips analyzed includes all enrolled. Number of hips demonstrating radiographic failure assessment at postoperative periods indicated is included in the outcome results posting. Number of hips available for evaluation is indicated in the results heading by postoperative period.
Measure: Number; unit: hips
Units Other Than Participants: Hips
Arm/Group | Trident® System | ABC System | Control
Number analyzed (Participants) | 177 | 166 | 87
Number analyzed (Hips) | 190 | 185 | 89
hips
  3 yr failure (160 Trident®/174 ABC/82 Control) | 0 | 0 | 0
  4 yr failure (153 Trident®/162 ABC/79 Control) | 0 | 0 | 0
  5 yr failure (128 Trident®/158 ABC/74 Control) | 0 | 0 | 0
  10 yr failure (60 Trident®/116 ABC/56 Control) | 0 | 0 | 0

4. Secondary Outcome: Hip Follow-Up Questionnaire
Description: A three question follow-up questionnaire was administered annually asking whether the participant is satisfied with the study total hip replacement(THR) (noted as "satisfied" below); whether they have any study hip pain (noted as "no pain" below); and whether they have had any surgery on the study hip during the previous year noted as "no surgery" below).
Time Frame: 6-10 years
Population: Participants may have one or both hips replaced. Number of participants/hips analyzed includes all enrolled. Number of hips with positive three question responses at postoperative periods indicated is included in the outcome results posting. Number of hips available for evaluation is indicated in the results heading by postoperative period.
Measure: Number; unit: hips
Units Other Than Participants: Hips
Arm/Group | Trident® System | ABC System | Control
Number analyzed (Participants) | 177 | 166 | 87
Number analyzed (Hips) | 190 | 185 | 89
hips
  6yr satisfied (Trident ®168/ABC 150/Control 79) | 163 | 146 | 76
  6yr no pain (Trident ®168/ABC 150/Control 79) | 142 | 129 | 63
  6yr no surgery (Trident ®168/ABC 150/Control 79) | 168 | 147 | 79
  7yr satisfied (Trident ®166/ABC 146/Control 71) | 161 | 145 | 71
  7 yr no pain (Trident ®166/ABC 146/Control 71) | 138 | 130 | 58
  7 yr no surgery (Trident® 166/ABC 146/Control 71) | 165 | 145 | 71
  8yr satisfied (Trident ®164/ABC 141/Control 75) | 160 | 141 | 73
  8yr no pain (Trident ®164/ABC 141/Control 75) | 140 | 127 | 68
  8yr no surgery (Trident ®164/ABC 141/Control 75) | 164 | 141 | 75
  9yr satisfied (Trident ®150/ABC 162/Control 83) | 148 | 161 | 83
  9yr no pain (Trident ®150/ABC 162/Control 83) | 128 | 150 | 73
  9yr no surgery (Trident ®150/ABC 162/Control 83) | 150 | 162 | 83
  10yr satisfied (Trident ®143/ABC 148/Control 76) | 142 | 148 | 76
  10yr no pain (Trident ®143/ABC 148/Control 76) | 123 | 136 | 65
  10yr no surgery (Trident ®143/ABC 148/Control 76) | 143 | 148 | 76
Statistical Analysis 1: Comparison: Trident® System vs ABC System vs Control; Compare the # of cases at 10 years satisfied with their total hip replacement for all three groups; Test type: Superiority or Other; p = 0.6011, Fisher Exact
Statistical Analysis 2: Comparison: Trident® System vs ABC System vs Control; Compare the # of cases at 10 years for having pain in their hip for all three groups; Test type: Superiority or Other; p = 0.2060, Fisher Exact

ADVERSE EVENTS:
Time Frame: 10 years
Description: Some participants were randomized to more than one hip system (17 participants/34 hips). Operative Site adverse events are reported by hip; systemic events are reported by participant. There were a total of 413 participants with 464 hips (190 Trident,185 ABC,89 Control) assessed.
Groups:
- Trident® System: Hips that received the Trident® Acetabular System with a ceramic insert and ceramic femoral head.
- ABC System: Hips that received the ABC Acetabular System with a ceramic insert and ceramic femoral head.
- Control: Hips that received the Omnifit Acetabular system with polyethylene insert and metal femoral head.
- All Participants: All participants combined.
Arm/Group | Trident® System | ABC System | Control | All Participants
Serious Adverse Events (participants affected / at risk) | 1/190 | 1/185 | 1/89 | 1/413
Other Adverse Events (participants affected / at risk) | 36/190 | 17/185 | 7/89 | 0/413
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Trident® System (N=190) | ABC System (N=185) | Control (N=89) | All Participants (N=413)
Non-operative Site Cardiac Disorders (Cardiac disorders) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 1 (1)
Operative Site Musculoskeletal and Connective Tissue Disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0/0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Trident® System (N=190) | ABC System (N=185) | Control (N=89) | All Participants (N=413)
Operative Site Musculoskeletal and Connective Tissue Disorder (Musculoskeletal and connective tissue disorders) | 36 (48) | 17 (17) | 7 (8) | 0/0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The disclosure restriction on the PI to publish results of this Clinical Study or the results of the activities hereunder, any abstract, manuscript, presentation or other communication shall be submitted to sponsor for review and approval at least 60 days prior to submission for publication. The sponsor retains the right to deny publication or, at its sole option, to revise the manuscript to delete proprietary or other confidential commercial information.